CLINICAL TRIAL: NCT05462288
Title: Entia Liberty: Home Study - Evaluation of Patient Preference for a Novel Full Blood Count Home Testing Device Versus Routine Venous Monitoring
Brief Title: Entia Liberty: Home Study
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 317614
Record Dates: First submitted 2022-06-20; First posted 2022-07-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group
  Interventions: Device: Entia Liberty

INTERVENTIONS:
Device: Entia Liberty — Home monitoring blood analyser

SUMMARY:
Participants will be testing with the home monitoring device over the course of their treatment. They are to self-test on days where they are due to be going into hospital for their routine pre-treatment blood tests. Participants will be asked to fill in interim questionnaires and a final questionnaire to answer the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Adequate English language skills (not requiring a translator) to participate in participant training and use the Liberty device
* Patients willing and able to perform capillary blood self-testing at the same frequency as routine full blood count monitoring
* Patients capable of providing informed consent before attending training
* Patients able to attend a 1-hour virtual training session within 2 weeks of joining the study
* Patients with a home Wi-Fi network or with adequate coverage at home via a 4G network
* Patients with access to a laptop or smartphone to facilitate training
* Patients with a diagnosis of ovarian or breast cancer
* Patients whose HCPs can confirm are undergoing systemic anti-cancer treatments within two weeks of enrolment, with treatment expected to continue for at least two cycles

Exclusion Criteria:

* Patients with haematological malignancies
* Patients with eyesight or hearing limitations or other disabilities that preclude the use of the Liberty device or participation in training unless they have a nominated caregiver who is capable of assisting with each test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New or existing patients on specific drug treatments recruited by their consultants
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
To assess patient preference for the Liberty self-testing pathway as compared to standard of care. | 12 months
  Patients will undergo the study procedures without change to their current pathway, at the end of the study, patients will compare the interventions via a SURVEY. The investigators will measure the success of the comparison by the % of patients who have chosen the investigators' product over the standard of care (4-5 rating out of 5).

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom